CLINICAL TRIAL: NCT04808817
Title: Assessment of Metabolic and Immune Profiles in Patients Receiving Immune Checkpoint Inhibitors (ICI) for Advanced Renal Cell Carcinoma or Lung Carcinoma.
Brief Title: Relationship Between Immunity and Metabolism in Patients Receiving Immune Checkpoint Inhibitors for Advanced Cancer. ( RIMEC )
Acronym: RIMEC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP201166; IDRCB 2020-A02262-37 (Other: ANSM)
Record Dates: First submitted 2021-03-08; First posted 2021-03-22 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Metabolism Disorder; Cancer; Immune Checkpoint Inhibitors
MeSH Terms: conditions — Metabolic Diseases; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients (Experimental)
  Interventions: Diagnostic Test: calorimetry, impedance measurement at baseline and after 3 months of treatment

INTERVENTIONS:
Diagnostic Test: calorimetry, impedance measurement at baseline and after 3 months of treatment — biobanking (30ml) for cytokines and complement dosages at baseline and after 3 months of treatment calorimetry and impedance measure will be collected at baseline and after 3 months of ICI treatment
  Other Names: biobanking (30ml)

SUMMARY:
Recent EMA and FDA approvals have made immune checkpoint inhibitors (ICI) a standard of care in cancer treatment. ICI, used alone or as a combination are now the backbone of renal cell and lung carcinoma treatment. However, a significant proportion of patients does not respond to ICI. Thus the identification of predictive response factor is a major issue.

While factors associated with the tumour and its micro environment have been widely studied, factors associated with the patient such as metabolism could also affect the response to ICI and remain poorly studied.

The hypothesis of the investigators is that dysmetabolims, via the induction of a chronic inflammatory state could induce a defect of lymphocyte production and activation as well as a modification of the immunogenicity of tumor cells and immune cells infiltration. The consequences could be a decrease in ICI response rate as well as an increase in immune related adverse events (irAEs).

To test this hypothesis, the investigators propose a prospective bi-centric exploratory study including 60 patients treated with ICI for advanced lung or renal cell carcinoma.

The data collected will be :

* Clinical (calorimetry, impedancemetry, survey of eating habits, tumour characteristics, epidemiological data),
* Biologics (baseline and 3-months plasma bio banking for standard biology, inflammation markers TNF- α, IL1-6-8-11-17, TGF-ß, TWEAK, complement study C3, C4, C4d, CH50, C1q, CD46)

Primary objective is to assess the response to ICI depending on metabolic status.

Secondary objectives are to study the relationships between metabolism / cytokines profile/ complement profile and ICI response.

The investigators seek to generate hypotheses and to obtain exploratory data before submission of a Hospital Clinical Research Program whose objective will be to evaluate the impact of dysmetabolism on overall survival and to characterize immune and anatomopathological profiles (using DNA microarrays and flow cytometry techinques) of patients treated with ICI for renal cell or lung carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥18 years
* patients receiving immune checkpoint inhibitors, used alone or as a combination with chemotherapy or tyrosine kinase inhibitor or other immune checkpoint inhibitor, for advanced renal cell or lung carcinoma.
* Patient Informed and signed the consent to participate in the research

Exclusion Criteria:

* patients with history of auto immune disease
* patients enrolled in an interventional study or be in the exclusion period following a previous research, if applicable
* Patient not affiliated to the social security scheme or under AME
* Patient under guardianship or curatorship or under legal protection
* Patient unable or unwilling to give written consent
* Pregnant patient

be in the exclusion period following a previous research, if applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-10-09 (Estimated)

PRIMARY OUTCOMES:
response rate according to metabolic status | 6 months from randomisation
  response rate after 6 months of ICI treatment (iRECIST criteria)

SECONDARY OUTCOMES:
6 months progression free survival according to metabolic status | 6 months from randomisation
  6 months progression free survival according to metabolic status
12 months overall survival according to metabolic status | 12months from randomisation
  12 months overall survival according to metabolic status
correlations between metabolism/ cytokines dosage/ complement dosage and response to ICI | 12 months from randomisation
  correlations between metabolism/ cytokines dosage/ complement dosage and
incidence of irAEs according to metabolic profile | 6 months from randomisation
  incidence of irAEs according to metabolic profile

CONTACTS AND LOCATIONS:
Overall Officials: SIMONAGGIO Audrey, MD, Principal Investigator — Hopital europeen Georges-Pompidou; Charles Vauchier, Principal Investigator — Hopital europeen Georges-Pompidou
Locations (2):
- France (2):
  - Hôpital Cochin, Paris, Île-de-France Region
  - AP-HP - Hôpital Européen Georges-Pompidou Paris, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Data sharing must respect the agreements made with funders.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).